CLINICAL TRIAL: NCT07100262
Title: Effect of Pulsed Electromagnetic Therapy on Chronic Dysphagia in Elderly Post-stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mostafa Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005715
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effortful swallow exercise (Active Comparator): The participants will receive two 30-minutes sessions of effortful swallow practice daily, 5 days/week, for 18 weeks.
  Interventions: Other: Effortful swallow exercise
- Pulsed electromagnetic therapy and effortful swallow exercise (Experimental): The participants will receive pulsed electromagnetic therapy for 30 minutes, 3 sessions weekly , in addition to two 30-minutes sessions of effortful swallow practice daily, 5 days/week, for 18 weeks.
  Interventions: Other: Effortful swallow exercise; Device: Pulsed electromagnetic therapy

INTERVENTIONS:
Other: Effortful swallow exercise — The participants will be practiced effortful swallow exercises as follows:
  When you are ready to swallow your saliva, squeeze your tongue against the roof of your mouth.
  B) As you swallow squeeze all the muscles in your throat. Imagine you are trying to swallow a large tablet or a golf ball.
  C) If it has been recommended by your speech and language therapist, this exercise may be repeated when eating and drinking.
  Frequency of exercise:
  Exercises will be two 30-minutes sessions of effortful swallow practice daily, 5 days/week.
  For every patient: 4 sets (1 set = 8-12 repetitions) 5 days/week, for 18 weeks.
Device: Pulsed electromagnetic therapy — The participants will receive pulsed electromagnetic therapy as the following:
  Position of patient: supine lying position with head supported by pillow. Sleeve of device: above anterior neck area.
  Parameters of application of device: according to programs for sarcopenia and muscular pain as the following:
  Power: 30 GAUSS. Frequency: in first 6weeks: 5Hz - second 6weeks: 10Hz - last 6weeks: 15Hz. Time of session: 30 min. Sessions frequency: 3 sessions per week. Time of treatment course: 18 weeks.
  Arms: Pulsed electromagnetic therapy and effortful swallow exercise

SUMMARY:
This study will be conducted to determine the effect of pulsed electromagnetic therapy on chronic dysphagia in elderly post-stroke Patients.

DETAILED DESCRIPTION:
Elders suffer from chronic dysphagia mainly after stroke (more than 6 months). Sarcopenia has been defined as a progressive and generalized disorder of skeletal muscle that involves accelerated loss of muscle mass and function. The prevalence of sarcopenia worldwide is up to 15% in healthy elderly, approximately 76% of acutely hospitalized elderly patients, and up to 69% of patients admitted for post-acute geriatric rehabilitation mainly post neurological stroke. This case series report is the first in the world scientific literature to demonstrate the effectiveness of Pulsed Electro Magnetic Frequency (PEMF) in gaining muscle strength and functionality in elderly sarcopenic patients. PEMF therapy, at least for the treatment of sarcopenia in the elderly, can be considered as the definitive evolution of electrical currents, with greater effectiveness and acceptance by the patient.

Skeletal muscle atrophy, a condition characterized by decreased muscle mass and contractility, is commonly observed in various pathological states, including prolonged inactivity, malnutrition and dysphagia. Findings examined in this trial suggest that antioxidants and Pulsed Magnetic Frequency (PMF) may alleviate impaired protein synthesis and degradation pathways in skeletal muscle atrophy. PMF showed a positive effect on the anabolic pathway.

A total of 26 studies were identified. Their intervention goals aimed to rehabilitate a broad spectrum of muscle groups within the oral cavity and pharynx and to improve the functions of swallowing, speech, facial expressions, or sleep breathing. Protocol duration ranged from 1 to 13 weeks, with various exercise repetitions (times per day) and frequency (days per week). Half of the studies reported using feedback to support the training, and these studies varied in the feedback strategy and technology tool. A total of 37 unique outcome measures were identified. Conclusions: This review demonstrated inconsistency across published studies in intervention goals and exercise protocols. It has also identified current limitations and provided recommendations for the selection of outcome measures while advancing a multidisciplinary view of oral and pharyngeal exercises in post-stroke recovery across relevant functions. The present study will examine effect of pulsed electromagnetic therapy on chronic dysphagia in elderly post stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients of both genders with chronic dysphagia.
* Their ages will be more than 65 years.
* Patients with body mass index (BMI) from 20kg/ m2 to 30kg/ m2.
* Patients had a stroke 6 months ago or more.
* Dysphagia symptoms started from the stroke time and continue till now.

Exclusion Criteria:

* Patients with anterior neck past surgeries, recent thoracic surgery and recent abdominal surgeries.
* Patients with neck tumors or traumatic lacerations on neck.
* Patients with cerebral hemorrhage affecting mainly oropharyngeal muscles.
* Patients with heart failure, myocardial infarction.
* Patients with any pulmonary diseases like plural effusion, pneumothorax, pulmonary fibrosis, emphysema.
* Cancer patients with or without metastasis.
* Patients with Alzheimer and Dementia.
* Blood pressure of less than 100/60 mmHg or more than 140/90 mmHg.
* Patients with psychological problems.
* Patients with psoriasis, burn and any dermatological problems in neck area.

Ages: 66 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Penetration Aspiration Score (PAS) | 18 weeks
  Standardized Fiberoptic Endoscopic Evaluation of Swallowing (FEES)will be applied for all subjects in both groups two times (before and after the trial), and PAS will be calculated. It is an 8-point ordinal scale, with 1 representing the least and 8 representing the highest or most severe score.
  1. Material does not enter airway.
  2. Material enters the airway, remains above the vocal folds, and is ejected from the airway.
  3. As point 2, but is not ejected from the airway.
  4. Material enters the airway, contacts the vocal folds, and is ejected from the airway.
  5. As point 4, but is not ejected from the airway.
  6. Material enters the airway, passes below the vocal folds, and is ejected into the larynx or out of the airway.
  7. Material enters the airway, passes below the vocal folds, and is not ejected from the trachea despite effort.
  8. Material enters the airway, passes below the vocal folds, and no effort is made to eject.
Eating Assessment Tool (EAT)-10 | 18 weeks
  It is a dysphagia screening tool developed to identify people at high risk of swallowing disorders. I twill be used for all subjects in both groups two times, the first before beginning of trial and the other after finishing the trial. it includes 10 items with 4 responses for each ranged from 0 to 4. 0 indicates no problem, and 4 indicates severe problem. Higher total score indicates more severity of the problem.
Functional Oral Intake Scale (FOIS): | 18 weeks
  It is a seven-point ordinal scale used to assess the functional ability of individuals with dysphagia to consume food and liquids orally. It was initially developed for stroke patients but is now widely used in adults and children with various neurological and other conditions affecting swallowing. The scale ranges from level 1 (no oral intake) to level 7 (total oral intake with no restrictions).
  Level 1: No oral intake. Level 2: Tube dependent with minimal or inconsistent oral intake. Level 3: Tube supplement with consistent oral intake. Level 4: Total oral intake of a single food consistency. Level 5: Total oral intake of multiple consistencies requiring special preparation.
  Level 6: Total oral intake of all consistencies with no special preparation. Level 7: Total oral intake with no restrictions.
Serum Creatinine/Cystatin C Ratio | 18 weeks
  Mindray Diluent Lyse device model BA88A will be used to assess Serum Creatinine/Cystatin C Ratio for all participants in both groups before and after treatment. It has been investigated as a potential marker for sarcopenia (age-related muscle loss). A typical range for the serum creatinine/cystatin C ratio might be between 6.45 and 24.14 for males and 4.62 and 23.49 for females. A higher ratio is associated with greater muscle mass, and lower ratios potentially linked to muscle loss.

CONTACTS AND LOCATIONS:
Overall Officials: Ayatallah Sheikhany, Professor, Study Director — Cairo University; Akram Sayed, Professor, Study Chair — Cairo University
Locations (1):
- Mohamed Ahmed Mostafa, Cairo, Egypt